CLINICAL TRIAL: NCT03518333
Title: Evaluation of the Tissue Genesis Icellator Cell Isolation System to Treat Erectile Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tissue Genesis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ED1002
Record Dates: First submitted 2018-04-24; First posted 2018-05-08 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, two-arm, blinded, randomized treatment. Covariate adaptive randomization will be used. Covariates included in the adaptive randomization process will be investigational center, history of diabetes, and radical prostatectomy.
Who Masked: Participant
Masking Description: Sham treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- ARM 1 (Experimental): Injection of adipose derived cells into penis followed six months later with sham control saline injection procedure
  Interventions: Device: Injection of adipose derived cells into penis
- ARM 2 (Experimental): Sham control saline injection procedure followed six months later by injection of adipose derived cells into penis
  Interventions: Device: Injection of adipose derived cells into penis

INTERVENTIONS:
Device: Injection of adipose derived cells into penis — Injection of Icellator-derived cells
  Other Names: Sham control intervention of injection of saline into penis

SUMMARY:
This clinical study is designed to investigate the safety and potential ability of relocated autologous SVF (stromal vascular fraction) to restore erectile function in men with ED (erectile dysfunction).

DETAILED DESCRIPTION:
Prospective, multi-center, two-arm, blinded, randomized treatment. Covariate adaptive randomization will be used. Covariates included in the adaptive randomization process will be investigational center, history of diabetes, and radical prostatectomy. The two randomized study arms are:

1. Treatment with SVF followed six months later with sham treatment (ARM 1)
2. Sham treatment followed six months later by treatment with SVF (ARM 2) Study population is 60 adult male subjects with organic erectile dysfunction (IIEF-EF score 11-22) of greater than 6 months' duration due to radical prostatectomy, diabetes mellitus, and/or vascular disease. Subjects will be followed for 12 months after initial treatment.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Chronic, organic ED, duration at least 0.5 years, with baseline IIEF-EF score of 11-22
* Willing to complete a 6-item erectile function questionnaire (IIEF-EF), a 4-week diary of sexual encounters (a single-item erection hardness assessment (EHS) and SEP-2 and SEP-3), 3 erectile function treatment Global Assessment Questions (GAQs), and 3 continence questions within 8 weeks before study treatment (baseline- except GAQs), and at each of the follow-up time points: 6 weeks (excluding EHS, SEP-2, SEP-3, and NPT), and 3, 6, 9, and 12 months after study treatment/ randomization
* Involved in a monogamous, heterosexual relationship for at least 3 months with both partners motivated to have or attempt sexual intercourse at least 4 times per month beginning two weeks after study treatment (subject reported)
* Willing to limit alcohol intake and eliminate use of recreational drugs for sexual encounters
* Willing to undergo two minor surgical procedure (small-volume liposuction, totaling approximately 60 - 120 cc) and two treatments of an injection of up to 30 cc of autologous SVF (or saline) into the corpora cavernosa over a 2- to 4-minute period, with a compression band applied at the base of the penis for total duration of up to 15 minutes
* Abdominal area amenable to two liposuction of at least 60-120 cc each of adipose tissue based on Investigator examination
* Mentally competent and able to understand all study requirements (based on investigator assessment)
* Willing to be available for all baseline, treatment and follow-up examinations required by protocol
* Willing to forego participation in any other study throughout the duration of this study unless receiving prior approval by Sponsor.

Exclusion Criteria:

* Evidence of prostate cancer which requires additional radiotherapy or other adjuvant therapy, or PSA > 0 after radical prostatectomy
* Previous pelvic or abdominal radiation therapy
* Anti-androgen therapy within the last 12 months or anti-androgen therapy of greater than 6 months in duration
* Untreated hypogonadism or low serum total testosterone (< 300 ng/dL)
* Clinically evident penile anatomical deformities (e.g., Peyronie's disease) or history of priapism
* Skin irritation, infection, wound, sore or disruption in the immediate areas of skin entry for abdominal liposuction or penile injection (including abdominal trauma and abdominal skin cancer (basal cell carcinoma, squamous cell carcinoma, and melanoma)
* Any previous penile implant or penile vascular surgery
* Current or previous malignancy other than localized prostate cancer or non-abdominal, non-melanoma skin cancer (successfully treated or treatable by curative excision or other local curative therapy- abdominal skin cancer is exclusionary)
* Uncontrolled hypertension or hypotension (systolic blood pressure > 170 or < 90 mm Hg, and diastolic blood pressure > 100 or < 50 mm Hg)
* Reported unstable cardiovascular disease (e.g., unstable angina, myocardial infarction within past 6 months, cardiac failure or life-threatening arrhythmia, congestive heart failure) or symptomatic postural hypotension within 6 months before screening
* Hemoglobin A1c > 10% within 8 weeks prior to study treatment
* Current urinary tract or bladder infection
* Drug, alcohol, anabolic steroid, or other substance abuse reported within the last year (subject reported)
* Subject's sexual partner is < 18 years of age, nursing, or known to be pregnant at screening, or wishes to become pregnant during the study period, or has any gynecologic problems, major medical conditions, or other factors that would limit participation in sexual intercourse to less than 4 times per month (subject reported)
* Weight less than 154 lbs/ 70 kg, or BMI ≥ 35
* Unable to limit or avoid NSAIDs for 15 days prior to treatment (subject reported)
* Bleeding or clotting disorder, use of anticoagulant therapy, or history of easy or excessive bruising
* Lab values for CBC, PT/PTT/INR, liver function and creatinine falling outside the normal lab values (see section 5.3 for further detail)
* Systemic autoimmune disorder
* Significant active systemic or localized infection
* Receiving immunosuppressant medications, including corticosteroids
* No prior regenerative medicine treatments or therapies
* Currently taking nitroglycerine (NTG) or other nitrate medication (such as isosorbide)
* Subjects who experience angina after taking PDE-5 inhibitors
* Any other condition, which, in the opinion of the Investigator, would contraindicate treatment, affect compliance, interfere with study evaluations, limit study participation, contraindicate sexual activity, or confound the interpretation of study results (e.g., clinical diagnosis of penile fibrosis, allergy to tumescence fluid or components of collagenase, cell therapy, change in alpha blocker drug therapy, sickle cell disease)

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult male subjects with organic erectile dysfunction (IIEF-EF score 11-22) of greater than 6 months' duration due to radical prostatectomy, diabetes mellitus, and/or vascular disease.
Enrollment: 60 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Objective: ability of adipose derived cells to restore erectile function using the 6-Item IIEF-EF score | 6 months
  Evaluate the ability of adipose derived cells to restore erectile function at 6 months using the 6-Item IIEF-EF score

SECONDARY OUTCOMES:
Safety Objective: assessment of any adverse events | 12 months
  Will be evaluated by the IDMC through assessment of any adverse events that occur during or after adipose tissue harvest and intracorporal injection of adipose derived cells through 12-month follow-up. All adverse events will be reviewed by the IDMC and the Sponsor at least every 3 months throughout enrollment, and at least annually throughout study follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Kosnik, PhD, Study Chair — Sponsor GmbH
Locations (5):
- United States (5):
  - San Diego Sexual Medicine, San Diego, California
  - James A. Simon, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Johns Hopkins Kimmel Cancer Center, Baltimore, Maryland
  - Scott Department of Urology, Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No